CLINICAL TRIAL: NCT03647904
Title: The SEMS Project: Staying Employed With MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Lauren Strober, Senior Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: E-944-16
Record Dates: First submitted 2018-01-25; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
Keywords: Employment; Self efficacy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Wait list control
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not know if individual were in the treatment group or waitlist control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEMS Project (Experimental): A comprehensive modular intervention consisting of wellness, fatigue management, cognitive remediation and psychological treatment. Treatment will consist of a total of 12 weeks.
  Interventions: Behavioral: SEMS Project
- Wait List Control (Other): Individuals in the wait list control arm will serve as controls for the first intervention group, but will receive the treatment following their three month assessment. The intervention following the waitlist control will be a comprehensive modular intervention consisting of wellness, fatigue management, cognitive remediation and psychological treatment. Treatment will consist of a total of 12 weeks.
  Interventions: Behavioral: SEMS Project

INTERVENTIONS:
Behavioral: SEMS Project — TThe intervention is a culmination of five empirically supported interventions: (1) The MS Wellness Program aimed at developing lifestyle strategies to enhance quality of living and cope with various aspects of MS; (2) The FACETS intervention, which aims to reduce fatigue and improve self-efficacy; (3) The Modified Story Memory technique, which improves new learning and memory; (4) The Speed of Processing training, which improves performance on measures of processing speed in persons with MS. Finally, the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders, a cognitive behavioral intervention, which improves psychological functioning and functional outcomes.

SUMMARY:
Description of Project: Multiple sclerosis (MS), a disorder of young and middle aged adults, is known to have a grave impact on one's well-being and incurs a significant cost to society due to the nearly 80% rate of unemployment. Over the past few decades, research has focused on increasing our understanding of the factors that lead to these high rates of unemployment in MS and ways to mitigate such factors. However, the majority of investigations examining the causes of unemployment in MS have been retrospective and limited their focus to factors such as demographics, disease severity and symptoms of MS (e.g., fatigue), and/ or work place features and accommodations. Few have examined the more intrinsic, or person-specific factors (e.g., personality, coping, health-related behaviors), which are also likely to significantly contribute to rates of unemployment in MS. In fact, these investigators have shown that personality characteristics, anxiety, depression, coping, and self-efficacy differ between individuals who are considering leaving the workforce and those staying employed; even in the presence of comparable demographics and disease variables. Based on these findings, and the knowledge that fatigue and cognition also greatly contribute to this decision, these investigators have proposed a comprehensive intervention that will target both the disease and person-specific factors in hope of assisting individuals with MS maintain their employment; the ultimate goal being to improve the overall quality of life and health of individuals with MS. The proposed modular intervention will be tailored to the individual based on a preliminary assessment and consist of cognitive rehabilitation, fatigue and symptom management, wellness intervention, psychological intervention, and occupational rehabilitation. Outcomes will be assessed following such intervention with the goal being either job maintenance or comparable life activities that will ensure continuity of purpose and satisfaction in life, health and health maintenance, and overall well-being.

DETAILED DESCRIPTION:
Multiple sclerosis (MS), a disorder of young and middle aged adults, has a grave impact on one's well-being and incurs a significant cost to society due to the nearly 80% rate of unemployment.1,2 Over the past few decades, research has focused on increasing our understanding of the factors that lead to the high unemployment rates in MS and ways to mitigate such factors. However, the majority of investigations examining the determinants of unemployment in MS have been retrospective and limited in their focus to factors such as demographics, disease symptoms and severity, and/or work place features and accommodations. Few have examined the more intrinsic, or person-specific factors (e.g., personality, coping, health-related behaviors), which are also likely to contribute to unemployment rates in MS. In fact, one of the earliest investigations examining the "common" factors associated with unemployment in MS asserted that premorbid personality, education level, quality of environment, and social/family network were likely to affect how an individual with MS reacted to their illness, including attitudes towards employment.2 By applying a new conceptual model that incorporates such person-specific factors, and controls for the more typical demographic and disease variable predictors of unemployment in persons with MS, these investigators have shown that personality characteristics, anxiety, depression, coping, and self-efficacy differ between individuals who are considering leaving the workforce and those who stay employed. Perhaps most striking, was the finding that these individuals had an average disease duration of only 6.7 years compared to 10.4 years of those staying employed. Moreover, 62% were within 5 years of diagnosis compared to only 36% among those staying employed. This nearly double rate may reflect poor adjustment to illness rather than a result of greater disability per se. Based on these findings, these investigators postulate that individuals who are considering leaving the workforce or reducing work hours could benefit from early intervention targeting person-specific vulnerability factors. Such intervention should not only address the cognitive, psychological, and physical consequences of MS, but also attend to vital premorbid and psychological factors (e.g., anxiety, coping, self-efficacy), which in some ways may better account for why individuals leave the workforce. Moreover, given the negative psychological and health consequences of unemployment, in general, it is imperative that we assist such individuals in maintaining their employment and adjustment to MS to ward of further reductions in overall well-being and quality of life. Thus, the proposed investigation aims to assist individuals with MS maintain their employment by developing a comprehensive intervention that will target both the disease and person-specific factors associated with unemployment in MS; the ultimate goal being to improve the overall quality of life and health of individuals with MS. The proposed modular intervention will be tailored to the individual based on a preliminary assessment, and it may consist of any or all relevant components of cognitive rehabilitation, fatigue and symptom management, wellness intervention, and psychological intervention. Outcomes will be assessed following such intervention, with the goal of enhancing greater commitment to work and job maintenance that will ensure continuity of purpose and satisfaction in life, health and health maintenance, and overall well-being. We will also assess change and process variables throughout the intervention to gain a better sense of the factors that facilitate change across these interventions. In sum, the specific aims of the proposed investigation are to:

Specific Aim 1: Develop and pilot a comprehensive and personally responsive (modular) intervention to assist individuals with MS remain in the workplace and examine the factors most associated with such change.

Specific Aim 2: Examine the immediate and long-term (3 month) outcomes of this intervention on functioning, well-being, self-efficacy, disease management, health, and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with MS based on McDonald Criteria

Exclusion Criteria:

* any neurological condition other than MS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Change in Work Commitment | baseline, immediate post-intervention, 3 month post-intervention
  One's ability to maintain their current work status and function as measured by the employment outcome questionnaire
Change in adjustment to MS | baseline, immediate post-intervention, 3 month post-intervention
  Self-reported perception of coping skills as measured by the COPE questionnaire
Change in self-efficacy | baseline, immediate post-intervention, 3 month post-intervention
  Self-reported self-efficacy as measured by the General Self-efficacy Questionnaire

SECONDARY OUTCOMES:
Change in mood | baseline, immediate post-intervention, 3 month post-intervention
  Self reported depression as measured by the Chicago Multiscale Depression Inventory questionnaire
Change in anxiety | baseline, immediate post-intervention, 3 month post-intervention
  Self-reported anxiety as measured by the State Trait Anxiety Inventory questionnaire
Change in psychological well-being | baseline, immediate post-intervention, 3 month post-intervention
  Self-reported psychological well-being as measured by the Ryff Psychological well-being scales
Changes in stress | baseline, immediate post-intervention, 3 month post-intervention
  Self-reported stress as measured by the Perceived Stress Scale questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Strober, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No